CLINICAL TRIAL: NCT04333654
Title: A Phase 1b, Randomized, Double-blinded, Placebo-controlled Study of Hydroxychloroquine in Outpatient Adults With COVID-19
Brief Title: Hydroxychloroquine in Outpatient Adults With COVID-19
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Rate of enrollment too slow to allow completion in a reasonable timeframe
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC16855; 2020-001269-35 (EudraCT Number); U1111-1249-6168 (Other: UTN)
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Coronavirus Infection
MeSH Terms: conditions — Coronavirus Infections | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydroxychloroquine (Experimental): Hydroxychloroquine, loading dose on day 1 followed by a daily maintenance dose during 9 days
  Interventions: Drug: Hydroxychloroquine SAR321068
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine SAR321068 — Pharmaceutical form:Tablet Route of administration: Oral
  Other Names: Plaquenil
  Arms: Hydroxychloroquine
Drug: Placebo — Pharmaceutical form:Tablet Route of administration: Oral
  Arms: Placebo

SUMMARY:
Primary Objective:

To assess the effect of hydroxychloroquine versus placebo on nasopharyngeal SARS-CoV-2 viral load in outpatient adults with COVID-19

Secondary Objectives:

* To assess the effect of hydroxychloroquine versus placebo on clinical signs and symptoms and progression of disease in outpatient adults with COVID-19
* To assess the safety and tolerability of hydroxychloroquine in outpatient adults with COVID-19

DETAILED DESCRIPTION:
The duration of the study per participant will be around 18 days (1 or 2 days of screening followed by a 10-day treatment period and a 4 to 6 days follow-up period)

ELIGIBILITY:
Inclusion criteria :

* Participants with diagnosis of COVID-19 via an approved or authorized molecular test
* Presence of symptoms compatible with COVID-19 at the time of screening
* Time between onset of symptoms and first dose of hydroxychloroquine or placebo is 96 hours or less
* Female participants must use an acceptable birth control method, as specified by each site and country

Exclusion criteria:

* COVID-19 disease requiring the use of supplemental oxygen
* Electrocardiogram (ECG) tracing with QTc interval > 450 ms for men, > 470 ms for women (Fridericia algorithm recommended)
* Bradycardia (< 50 beats/min)
* History of cardiac disease (eg. congestive heart failure, myocardial infarction)
* History of Glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Women who are pregnant or breastfeeding
* Concurrent antimicrobial therapy
* Known hypersensitivity to hydroxychloroquine or other 4-aminoquinoline compounds
* Hydroxychloroquine use within 2 months before enrollment
* History of severe skin reactions such as Sevens-Johnson syndrome and toxic epidermal necrolysis
* History of retinopathy
* History of arrythmia, concurrent use of anti-arrhythmic drugs, or family history of sudden cardiac death
* History of severe renal disease (treatment with dialysis or phosphate binders) or hepatic impairment

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-04-12 (Actual); Primary Completion 2020-05-26 (Actual); Study Completion 2020-05-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Day 3 in nasopharyngeal SARS-CoV-2 viral load (if quantitative PCR is available) | Baseline to Day 3
  Viral load assessed by PCR from a nasopharyngeal swab
Number of participants by PCR result status (positive or negative) (if quantitative PCR is not available) | Baseline to Day 3
  Viral load assessed by PCR from a nasopharyngeal swab - 2. Viral load assessed by PCR from a nasopharyngeal swab

SECONDARY OUTCOMES:
Change from baseline to Day 5 in nasopharyngeal SARS-CoV-2 viral load | Baseline to Day 5
  Viral load assessed by PCR from a nasopharyngeal swab
Number of participants by PCR result status (positive or negative) | Baseline to end of study (Day14)
  Viral load assessed by PCR from a nasopharyngeal swab
Number of participants with COVID-19 symptoms by severity | Baseline to end of study (Day14)
  COVID-19 symptoms (feverishness, sore throat, cough, shortness of breath, myalgias) will be scored by the participant on a 4-point scale ( 0 =none; 1 = mild; 2 = moderate; 3 = severe)
Time to resolution of COVID-19 Symptoms | Baseline to end of study (Day14)
  COVID-19 symptoms (feverishness, sore throat, cough, shortness of breath, myalgias) will be scored by the participant on a 4-point scale ( 0 =none; 1 = mild; 2 = moderate; 3 = severe). Resolution of a symptom is defined as when a symptom previously scored ≥ 1 on the scale is scored as 0
Time to resolution of fever | Baseline to end of study (Day14)
  Resolution of fever defined as the first day of 2 consecutive daily temperatures < 37.7 C
Percentage of participants with resolution of fever | Baseline to end of study (Day14)
  Resolution of fever defined as the first day of 2 consecutive daily temperatures < 37.7 C
Percentage of participants hospitalized | Baseline to end of study (Day14)
Number of participants with Adverse Events | Baseline to end of study (Day14)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (7):
- Investigational Site Number 8400001, Boston, Massachusetts, United States
- Belgium (2):
  - Investigational Site Number 0561001, Brussels
  - Investigational Site Number 0561002, Lodelinsart
- France (2):
  - Investigational Site Number 2501001, Bordeaux
  - Investigational Site Number 2501002, Paris
- Netherlands (2):
  - Investigational Site Number 5281001, Groningen
  - Investigational Site Number 5281002, Harderwijk

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: EFC16855 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25258&tenant=MT_SNY_9011